CLINICAL TRIAL: NCT04243187
Title: Evaluation of Gastrointestinal Symptoms Following Chilean Native Beans Consumption
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Natalia Jara (Other)
Collaborators: Instituto de Nutrición y Tecnología de los Alimentos (Other)
Responsible Party: Sponsor-Investigator, Natalia Jara, MD Msc, University of Chile
Organization: University of Chile (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Porotos
Record Dates: First submitted 2020-01-23; First posted 2020-01-28 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Gastrointestinal Disease; Flatulence; Gastrointestinal Tolerance; Distension; Bowel; Bloating
Keywords: phaseolus; symptoms; expired hydrogen; bloating; bean; tolerance; beans
MeSH Terms: conditions — Gastrointestinal Diseases; Flatulence; Dilatation, Pathologic; Spinocerebellar Ataxia 31

STUDY DESIGN:
Intervention Model Description: 10 subjects, 8 visits, once a week, for bean intake (80 grams of dried beans, soaked for 12 hours, cooked in new water for 1.5 - 2 hours. This is approximately 160 grams of cooked beans).
  Four varieties of beans (3 native and 1 commercial) will be analyzed, which will be consumed by duplicate for participants (8 visits).
  A ninth visit will be made to perform a exhaled hydrogen test with raffinose (5 grams), as a positive control.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Clinical Study (Experimental): 9 visits, once a week, for bean intake (80 grams of dried beans, soaked for 12 hours, cooked in new water for 1.5 - 2 hours. This is approximately 160 grams of cooked beans).
  Four varieties of beans (3 native and 1 commercial) will be analyzed, which will be consumed in duplicate by participants (8 visits).
  A ninth visit will be made to perform a exhaled hydrogen test with raffinose (5 grams), as a positive control.
  Interventions: Other: Chilean Native Beans

INTERVENTIONS:
Other: Chilean Native Beans — In each visit the participant would have to:
  1. Fill a survey of gastrointestinal symptoms and basal bowel movements ("THE GASTROINTESTINAL SYMPTOM RATING SCALE (GSRS))
  2. Fill a survey of food consumption
  3. Bean plate intake
  4. Expired hydrogen test, which consists of exhaling air in a syringe every 20 minutes for 12 times (4 hours in total). During this time the participant can do quiet activities (not physical activity).
  5. Fill surveys of gastrointestinal symptoms (online or on paper), during the hydrogen test, at 12 and 24 hours (3 times). During this time (1 day before and 2 days later) the participant cannot eat other bloating foods (legumes, cauliflower, broccoli, lettuce, cabbage, artichokes, onions, topinambur and others described in the food survey).

SUMMARY:
The oligosaccharide content (raffinose, stachyose, and verbascose) in legumes would be responsible for gastrointestinal symptoms (bloating, pain, meteorism), associated with its consumption.

We would evaluate consumption of 3 varieties of chilean native beans, and evaluate gastrointestinal symptoms produced along with expired H2 test, to correlate this with the amount of oligosaccharide content.

DETAILED DESCRIPTION:
Different varieties of legumes have different oligosaccharide contents, in a study in Poland, it is described that the content of stachyose between 3 varieties can be as different as 493 mg, 865 mg or 1200 mg per 100 grams of dried beans (Slupski 2014). Along with this it has been described that the different culinary preparations of the legumes decrease the anti-nutritional factors, so, when soaking for 6 hours it shows 16.5% of undigested sugars reaching the small intestine, but it is possible to digest 95% in the colon (Noah 1998). Soaking for 16 hours, decreases 85% phytate content, 84% tannin content, 25% raffinose content, 25% stachyose and 41% verbascose (Hurtado 2001).

The oligosaccharide content (raffinose, stachyose, and verbascose) would be responsible for gastrointestinal symptoms (bloating, pain, meteorism), associated with legume consumption.

This is because these sugars are galactooligosaccharides, which are not digested in the human intestine because it does not have an alpha-galactosidase enzyme (Hessels 2003).

In our study, 25 varieties of Chilean bean are being evaluated, with nutritional analysis, resulting in a variation between 18 and 25 grams of protein per 100 grams dry (unpublished data), the oligosaccharide content still pending will be evaluated for Select the 3 varieties that contain more proteins and less oligosaccharides.

These varieties with better nutritional "profile" will be selected, to be evaluated clinically.

ELIGIBILITY:
Inclusion Criteria:

* Beans consumption on a regular basis (at least once a week)
* Without obvious intolerance to beans intake

Exclusion Criteria:

* Clinical history of recurrent gastrointestinal discomfort
* Diagnosis of any gastrointestinal disease (gastroesophageal reflux, gastritis, irritable bowel syndrome, chronic diarrheal syndrome, etc.).
* Meeting Rome IV criteria for diagnosis of irritable bowel syndrome.
* Use of medications that affect gastrointestinal motility (omeprazole, metoclopramide, domperidone, loperamide, etc.) or antibiotics in the last month.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-04-01 (Estimated); Primary Completion 2020-07-31 (Estimated); Study Completion 2020-10-31 (Estimated)

PRIMARY OUTCOMES:
Gastrointestinal symptoms | 4 months
  We will evaluate the difference in the THE GASTROINTESTINAL SYMPTOM RATING SCALE (GSRS), with the intake of different native beans
Gastrointestinal symptoms | 4 months
  We will evaluate the difference in the "bristol stool chart" with the intake of different native beans

SECONDARY OUTCOMES:
Exhaled Hydrogen Test | 4 months
  We will evaluate the difference in the exhaled hydrogen test with the intake of different native beans

IPD SHARING:
Plan to Share IPD: Yes
De-identified data for all participants will be available
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 6 month after completion of the study
Access Criteria: data access requests will we analyzed by the principal investigator.